CLINICAL TRIAL: NCT04090203
Title: Boiled Peanut Oral Immunotherapy for the Treatment of Peanut Allergic Pediatric Patients
Brief Title: Boiled Peanut Oral Immunotherapy
Acronym: BPOIT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alton Melton (Other)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor-Investigator, Alton Melton, Sponsor-Investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPOIT 18-1294
Record Dates: First submitted 2019-05-30; First posted 2019-09-16 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Peanut Hypersensitivity
Keywords: Peanut; Allergy
MeSH Terms: conditions — Peanut Hypersensitivity; Hypersensitivity | interventions — Immunotherapy

STUDY DESIGN:
Intervention Model Description: Prospective open label phase I
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Boiled Peanut Powder (Experimental): Boiled Peanut Powder
  Interventions: Drug: Boiled Peanut Powder

INTERVENTIONS:
Drug: Boiled Peanut Powder — Oral Immunotherapy will be administered utilizing a powder derived from boiled peanuts. Treatment will begin with an initial escalation day in which dosing is begun at 0.1 mg peanut protein and escalated to a final dose of 6 mg peanut protein. Doses are ingested orally. The subjects will continue daily oral ingestion of doses at home and return for updosing every 2 weeks to a final maintenance dose of 300 mg peanut protein. The subjects will continue daily oral ingestion of the peanut product for a minimum duration of 28 days before undergoing exit DBPCFC. At the conclusion of the study, patients will be offered continued maintenance therapy off study in line with current specialty standards.
  Other Names: Immunotherapy

SUMMARY:
Prospective Phase 1 clinical trial providing proof of concept data on boiled peanut oral immunotherapy (OIT) for the treatment of peanut allergy in children. The investigators hypothesize that the proportion of subjects successfully desensitized with boiled peanut OIT is greater than the theoretical placebo rate of 20%.

DETAILED DESCRIPTION:
Oral Immunotherapy will be administered utilizing a powder derived from boiled peanuts. Treatment will begin with an initial escalation day in which dosing is begun at 0.1 mg peanut protein and escalated to a final dose of 6 mg peanut protein. Doses are ingested orally. Participants will continue daily oral ingestion of doses at home and return for updosing every 2 weeks to a final maintenance dose of 300 mg peanut protein. Participants will continue daily oral ingestion of the peanut product for a minimum duration of 28 days before undergoing exit double blind placebo controlled food challenge. At the conclusion of the study, participants will be offered continued maintenance therapy off study in line with current specialty standards.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-16 years
* History of immediate hypersensitivity reaction to peanut
* Evidence of IgE mediated peanut hypersensitivity within a 12 month period of study enrollment
* SPT with wheal/flare of at least 3 x 6 mm and/or Peanut specific IgE >0.35 kU/L

Exclusion Criteria:

* History of life threatening peanut anaphylaxis
* Asthma requiring more than medium dose ICS
* Prior participation in oral immunotherapy, sublingual immunotherapy or epicutaneous immunotherapy
* Oat allergy
* Cardiovascular Disease
* Use of beta-blockers (oral), angiotensin converting enzyme inhibitors, angiotensin receptor blockers, or calcium channel blockers
* Use of steroid medications in the following manners:
* Daily oral steroid dosing for greater than 1 month during the past year
* Burst or steroid course in the past 3 month before inclusion
* Greater than 2 bursts oral steroid courses in the past year of at least 1 week duration
* Pregnancy or lactation
* Eosinophilic Gastrointestinal Disease
* History of food protein-induced enterocolitis
* History of developmental delay or speech delay that precludes age- appropriate communication, in the opinion of the investigator

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaclyn Bjelac, MD, Principal Investigator — Staff
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Boiled Peanut Powder
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Boiled Peanut Powder
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 4 [1 to 12]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Increase in Tolerance to Peanut in Pediatric Patients With Peanut Hypersensitivity Reported as the Percentage of Participants Successfully Desensitized.
Description: The percentage of patients able to consume a single dose of 300 mg or greater of peanut protein with no dose limiting symptoms at exit food challenge are considered 'successfully desensitized'. Any enrolled participants who did not tolerate the 300 mg dose or did not complete the exit food challenge for any reason are considered not successfully desensitized. The percentage of successfully desensitized participants is presented with corresponding lower bound of the one-sided 95% CI, calculated as the lower bound of a two-sided 90% exact confidence interval.
Time Frame: 18 weeks
Population: All participants who enrolled in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Boiled Peanut Powder
Number analyzed (Participants) | 8
percentage of participants | 75 [40 to 100]
Statistical Analysis 1: Comparison: Boiled Peanut Powder; The null hypothesis was that the percentage of patients who were successfully desensitized was less than or equal to 20%, and the alternative hypothesis was that this percentage was greater than 20%. Assuming 80% of study participants would be successfully desensitized, a sample size of 10 patients would provide greater than 90% power to reject the null hypothesis using a one-sided exact binomial test with a significance level of 0.05; Test type: Superiority; p = 0.001, Exact binomial test — The test was performed at a one-sided significance level of 0.05; The null hypothesis of the exact binomial test was that the percentage of patients who were successfully desensitized was less than or equal to 20%; Percentage = 75.0, 95% CI 1-sided [lower limit 40.0] — The percentage of successfully desensitized participants is presented with a one-sided 95% CI, obtained from the lower bound of the two-sided 90% Clopper-Pearson exact confidence interval

ADVERSE EVENTS:
Time Frame: All reportable events will be recorded with start dates occurring any time after informed consent is obtained until 7 days (for non-serious AEs) or 30 days (for SAEs) after the last day of study participation. Study participation could last for a maximum of up to 35 weeks.
Arm/Group | Boiled Peanut Powder
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 2/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Boiled Peanut Powder (N=8)
Anaphylaxis - Hives; redness and swelling of eyes; cough; difficulty breathing (Immune system disorders) | 1 (1)
Coughing and wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Globus sensation; audible change in voice; dysphagia (Immune system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Boiled Peanut Powder (N=8)
Abdominal Pain (Gastrointestinal disorders) | 3 (9)
Abdominal Pain, Diarrhea (Gastrointestinal disorders) | 1 (1)
Abdominal Pain, Facial Flushing, Head Pain, Pruritus, Malaise (Immune system disorders) | 1 (1)
Abdominal Pain, Non-Cardiac Chest Pain (Gastrointestinal disorders) | 1 (1)
Abdominal Pain, Upset Stomach, Reflux (Gastrointestinal disorders) | 1 (1)
Belching (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough, Urticaria, Lip/Mouth Pruritus, Vomiting (Immune system disorders) | 1 (1)
Cough, Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 2 (8)
Eczema, Pruritus (Immune system disorders) | 1 (1)
Eczema, Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Eyelid Dysfunction (Redness/Swelling) (Skin and subcutaneous tissue disorders) | 1 (1)
Facial Rash, Mucositis Oral (Immune system disorders) | 1 (1)
Fever, Vomiting (Infections and infestations) | 1 (1)
Gastrointestinal Pain (Gastrointestinal disorders) | 1 (1)
Lip/Mouth Pruritus (Immune system disorders) | 1 (48)
Lip/Mouth Pruritus, Abdominal Pain, Throat Pruritus (Immune system disorders) | 1 (1)
Lip/Mouth Pruritus, Eye Pruritus, Vomiting (Immune system disorders) | 1 (1)
Lip/Mouth Pruritus, Nausea (Immune system disorders) | 1 (1)
Lip/Mouth Pruritus, Rash Maculo-Papular (Immune system disorders) | 1 (1)
Lip/Mouth Pruritus, Throat Pruritus (Immune system disorders) | 1 (2)
Lip/Mouth Pruritus, Throat Pruritus, Nausea (Immune system disorders) | 1 (1)
Nasal Congestion, Urticaria (Immune system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (6)
Pruritus (Immune system disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Pruritus, Cough (Immune system disorders) | 1 (1)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis (General disorders) | 1 (1)
Rhinitis, Nasal Congestion (General disorders) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Serous Otitis (Ear and labyrinth disorders) | 1 (1)
Throat Pruritus (Immune system disorders) | 1 (11)
Urticaria (Immune system disorders) | 2 (2)
Urticaria, Cough (Immune system disorders) | 1 (2)
Urticaria, Eye Pruritus, Nasal Congestion (Immune system disorders) | 1 (1)
Urticaria, Periorbital Edema (Immune system disorders) | 1 (1)
Urticaria, Rash Maculo-Papular (Immune system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (7)
Vomiting, Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Vomiting, Nasal Congestion, Chest Wall Pain (Gastrointestinal disorders) | 1 (1)
Vomiting, Urticaria (Immune system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Enrollment was paused due to institutional IRB regulations during the COVID-19 pandemic. After resumption of enrollment, the study proceeded as planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2020-02-12): https://cdn.clinicaltrials.gov/large-docs/03/NCT04090203/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/03/NCT04090203/SAP_001.pdf
  • Informed Consent Form (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/03/NCT04090203/ICF_002.pdf